CLINICAL TRIAL: NCT04188145
Title: A Randomized Phase III Study Comparing Maintenance Treatment With Fluoropyrimidine + Bevacizumab Versus Fluoropyrimidine After Induction Chemotherapy for a Metastatic Colorectal Cancer
Acronym: BEVAMAINT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 71
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoropyrimidine (Active Comparator)
  Interventions: Drug: Fluoropyrimidine
- Fluoropyrimidine + Bevacizumab (Active Comparator)
  Interventions: Drug: Fluoropyrimidine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fluoropyrimidine — Option 1: Capecitabine 1250 mg/m2 twice daily (i.e. 2500 mg/m²/d) (D1 to D14, D1 = D22) For frail patients according to investigator evaluation capecitabine dose may be reduced to 1000 mg/m2 twice daily (2000 mg/m²/d).
  Or Option 2: Capecitabine 625 mg/m2 twice daily (i.e. 1250 mg/m²/d) (D1 to D21, D1 = D22) Or Option 3: LV5FU2 simplified (folinic acid 200 mg/m² (or Elvorin 400 mg/m²) IV during 2h followed by 5-FU bolus IV of 400 mg/m² during 10 min and IV continuous 5-FU at 2400 mg/m² during 46h). (D1=D15).
Drug: Bevacizumab — Option 1 and Option 2 : D1 bevacizumab 7.5 mg/kg IV (D1=D21). See smPCs for infusion time of bevacizumab.
  Or Option 3: D1 bevacizumab 5 mg/kg IV (D1=D15). See smPCs for infusion time of bevacizumab
  Arms: Fluoropyrimidine + Bevacizumab

SUMMARY:
The aim of BEVAMAINT is to improve benefic effect of maintenance therapy after a first line of induction chemotherapy for patients with colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma before induction treatment
* Measurable or non-measurable lesion before the induction treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Metastatic, unresectable disease according local practice after induction treatment
* ECOG performance status ≤ 2
* Disease control (complete response, partial response or stable disease) after 4-6 months of frontline induction chemotherapy with doublet (fluoropyrimidine + irinotecan or oxaliplatin) or triplet (fluoropyrimidine + irinotecan + oxaliplatin) +/- (cetuximab, panitumumab, bevacizumab) or IAH chemotherapy
* Life expectancy > 3 months
* Age ≥ 18 years
* Patient is at least 4 weeks from any major surgery
* Total bilirubin < 25 µmol/L, ASAT < 3 x ULN, ALAT < 3 x ULN (ASAT , ALAT < 5 x ULN in case of hepatic metastasis) , PT >60% , PAL<2.5 x ULN ( < 5 x ULN in case of hepatic metastasis) - Neutrophils > 1500/mm3, platelets > 100 000/mm3, haemoglobin ≥ 9 g/dL
* Creatinin clearance > 30 ml/min (MDRD) - if creatinin clearance comprised between 30 and 50 ml/min, see smPCs for dose adjustments
* Proteinuria ≤ 2+ (dipstick urinalysis) (if more than 2+, so proteinuria at or ≤1g/24hour must be ≤1g)
* Patient is able to understand, sign, and date the written informed consent
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for premenopausal female patients
* Male and female patients of childbearing potential agree to use a highly effective contraceptive measure
* Patient affiliated to a social security system

Exclusion Criteria:

* Myocardial infarction, severe coronaropathy or severe cardiac dysfunction less than 6 months prior randomization
* Follow-up impossible
* Patients with all metastases resected (R0/R1) after induction chemotherapy
* Patient with a hand-foot syndrome > 1 before maintenance treatment
* Known brain or leptomeningeal metastases
* Other concomitant or previous malignancy, except: adequately treated in situ carcinoma in complete remission for > 5 years
* Uncontrolled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy
* Pregnancy or breast feeding
* Treatment with sorivudine or analogs (brivudine)
* Treatment with phenytoin or analogs
* Partial or complete DPD deficiency (Uracilemia ≥ 16 ng/ml)
* Peptic ulcer not healed after treatment
* Any contraindication to bevacizumab or fluoropyrimidine treatments according to the updated SmPC
* Intestinal perforation or intestinal fistula
* Previous or active gastrointestinal bleeding
* Thromboembolic event and/or history of thromboembolic event
* Severe hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Time-to-Treatment Failure (TTF) | 8 months
  Will be calculated from date of randomization (after the end of induction chemotherapy) to first radiological progression (according to RECIST 1.1) or death or start of a new chemotherapy (induction regimen or second line) or end of maintenance treatment without further chemotherapy, even if there is no radiological progression. Patients alive with no radiological progression and under maintenance treatment will be censored at the date of last news.

SECONDARY OUTCOMES:
Progression-free survival (PFS1) | 16 months
  Defined as the time between randomization and the first radiological progression (according to RECIST 1.1) or death (whatever occurs first). Patients alive and without progression will be censored at the date of last news.
Progression-free survival (PFS2) | 16 months
  Defined as the time between the end of maintenance treatment (whatever the reason is) and the radiological progression after this end of maintenance treatment or death whatever the cause. Patients alive and without progression will be censored at the date of last news.
Overall Survival (OS) | 3 years
  Defined as the time between randomization and death (any cause). Patients alive will be censored at the date of last news.
Safety | 3 years
  Toxicities will be graded according to the NCI-CTC v 4.0 criteria before each cycle.
Quality of Life (QoL) | 3 years
  Assessed at each evaluation with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France